CLINICAL TRIAL: NCT03591718
Title: A Phase I, Blinded Within Dose Groups, Multiple Dose, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Different Titration Schemes of BI 456906 in Patients With Obesity and Overweight.
Brief Title: A Study to Test Different Doses of BI 456906 in Patients With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1404-0003; 2018-000250-22 (EudraCT Number)
Record Dates: First submitted 2018-07-04; First posted 2018-07-19 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 456906 (Experimental)
  Interventions: Drug: BI 456906
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 456906 — Solution for injection
  Arms: BI 456906
Drug: Placebo — solution for injection
  Arms: Placebo

SUMMARY:
Main objective is to investigate the tolerability of different titration schemes of BI 456906 in otherwise healthy patients with obesity/overweight, and to determine a titration scheme for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years and < 70 years of age at screening
* Body Mass Index (BMI) ≥ 27 kg/m2 and <40 kg/m2 at screening
* A minimum absolute body weight of 70 kg at screening and a stable body weight (defined as no more than 5% change) 3 months prior to screening
* HbA1c <6.5%
* Further inclusion criteria apply

Exclusion Criteria:

* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Supine blood pressure (BP) ≥160/100 mmHg at screening
* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomization or planned within 12 months after screening
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Further exclusion criteria apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Cumulative number [N (%)] of patients withdrawn from up-titration by up-titration scheme | Up to 132 days

SECONDARY OUTCOMES:
AUC0-168 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 168h) | Up to 168 hours
Cmax (maximum measured concentration of the analyte in plasma) after first dose | Up to 132 days

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Profil Mainz GmbH & Co. KG, Mainz
  - Profil Institut für Stoffwechselforschung GmbH, Neuss

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. Studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. Studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to: 1.find information in order to request access to clinical study data, for listed studies. 2.request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement'.

REFERENCES:
- [Derived] Jungnik A, Arrubla Martinez J, Plum-Morschel L, Kapitza C, Lamers D, Thamer C, Scholch C, Desch M, Hennige AM. Phase I studies of the safety, tolerability, pharmacokinetics and pharmacodynamics of the dual glucagon receptor/glucagon-like peptide-1 receptor agonist BI 456906. Diabetes Obes Metab. 2023 Apr;25(4):1011-1023. doi: 10.1111/dom.14948. Epub 2023 Jan 30. PMID 36527386
- See also: Related Info — http://www.mystudywindow.com